## Sensory Integration of Auditory and Visual Cues in Diverse Contexts Statistical Analysis Plan June 1<sup>st</sup>, 2020 NCT04479761

For each of measure of interest and for each environment (stars, subway), we will fit a linear mixed effects model. Each model will include main effects of group, visual condition, and auditory condition, as well as all two and three-way interactions. The models will also control for age. For aim 1, we will assess the significance of contrasts between no sounds / dynamic sounds for the different visual conditions and groups. For aim 2, the same will be done for contrasts between no sounds / static sounds. These models estimate the difference in visual weighting and reweighting between the groups, maximizing the information we can obtain from the data by accounting for the inherent multilevel study design (person, conditions, repetitions). Since each person completes various trials for each condition, the linear mixed effects model accounts for these sources of variability.<sup>81</sup> *P*-values for the fixed effects will be calculated using the Satterthwaite approximation for the degrees of freedom for the T-distribution<sup>82</sup>.